CLINICAL TRIAL: NCT03026101
Title: Understanding the Role of the External Carotid Artery in the Pathophysiology of Migraine Pain
Brief Title: Understanding the Pathophysiology of Migraine Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-8335
Record Dates: First submitted 2016-12-27; First posted 2017-01-20 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Migraine Disorders; Migraine, Classic; Migraine Without Aura
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Migraine Intervention (Experimental): A catheter will be placed in the symptomatic side external carotid artery and a diagnostic angiogram will be performed. The diameter of the occipital artery, superficial temporal artery and middle meningeal artery will be measured. Depending on the location of the headache superselective catheterization with microcatheter will be placed in either superficial temporal artery, occipital artery or middle meningeal artery. A volume of 50µg of nitroglycerin diluted in 10ml saline will be injected into the branch of interest dependent on laterality and location of symptoms over 30 seconds, to be delivered into these vessels only. 1 minute after superselective nitroglycerin injection the patient will be questioned as to whether the headache has been induced. A follow up diagnostic angiogram of the external carotid artery will be performed 3 minutes after injection. If there is no response to the lower 50µg, a dose of 150µg nitroglycerin in 10ml saline will be administered.
  Interventions: Other: Nitroglycerin

INTERVENTIONS:
Other: Nitroglycerin — Intra-arterial adminstration to dilate external carotid artery branches to replicate migraine pain
  Other Names: Nitrostat

SUMMARY:
Migraine is the most common headache disorder, prevalent in 18% of females and 6% of males. Emergency room visits, physician consults, hospitalizations, medications, and indirect costs such as lost work days and decreased productivity place the global economic burden of migraines at over 20 billion dollars. It is prevalent in 28 million people in the US alone. Symptoms include unilateral, throbbing, debilitating headache pain accompanied by nausea, vomiting, photophobia, and phonophobia. Upwards of 75% of migraine patients have reduced functionability, have lost time at work, and 1/3 of patients require bed rest to manage the symptoms. The health-related impact on quality of life was comparable with that experienced by patients with congestive heart failure, hypertension, or diabetes.

While the burden of migraines on our society is clear, the pathophysiology of migraines remains largely unknown. The trigeminovascular system, including the external and internal carotid arteries and their associated sensory fibers which subserve the head have long been implicated in the pain and cutaneous allodynia experienced by migraine patients. Wolff in 1953, was the first to posit that migraine headache pain is the caused by dilation or circumferential expansion of the extracranial carotid artery. He demonstrated that migraineurs had twice the pulse amplitude in their external carotid arteries compared to control subjects and these changes were directly correlated to migraine symptoms. In a 2008 study, randomized migraineurs received nitroglycerin via peripheral IV or placebo for 20 minutes prior to obtaining magnetic resonance angiography (MRA). Nitroglycerin, a potent dilator of blood vessels, reliably induced migraine-like pain in up to 80% of patients, and transient dilation of vessels of up to nearly 40%, mostly in the extracranial vessels. Sumatriptan's efficacy in migraine relief provides further evidence for this theory, as it is a selective extracranial vessel constrictor which does not cross the blood brain barrier.

The goal of this current work is to utilize the direct, real-time angiography, which provides a high resolution map of vasculature, and demonstrate changes in vessel flow in patients who have migraine headache attacks. This information may guide therapeutic interventions in the future in order to better treat these migraine patients.

DETAILED DESCRIPTION:
The goals of the current study will be to demonstrate time-linked headache pain after super-selectively administration of vasodilatory medications to external carotid artery branches, and then observe vessel changes and presumed headache relief with transient occlusion of the same vessel. This work will be the first study to attempt to correlate the onset of headache pain with selective vessel dilation as seen on angiography, which has spatial and temporal resolution far superior to MRA imaging. It will also test the effect of transient vessel occlusion in this setting for possible relief of symptoms. This novel approach to migraine evaluation could advance the understanding of the disorder and steer future research towards more effective management of migraine pain. Only patients who have failed all medical and non-invasive therapies will be considered for this study.

Subjects will be evaluated by history and physical during a clinic visit for their migraines and the 'pre-angiography' screening will be performed at that time. A thorough history of their migraine symptomatology, if they agree to participate, will be obtained via questionnaire, including: severity, location, quality, alleviating and exacerbating symptoms, medications used, associated symptoms, frequency, and degree of debilitation. This information will be collected regarding their migraines uniquely for this study. The patients will also be given a headache log with each one of these measures as a column with space in each row to describe individual migraine episodes between their first clinic visit and their angiogram date. After this clinic visit, they will be scheduled for angiography between 2 and 4 weeks for the evaluation of their migraines. Their headache logs will be collected prior to their procedures.

The main portion of this study will occur during a single angiography session and the following 5 hours post-procedure period during which the patient will be monitored closely as part of standard post-angiogram care. An anesthesiologist will be present throughout the procedure and available for medication review and administration as needed. The patients will sign a consent form at the start of the day and will be reminded that they have the option of not participating in the study and continuing their normal migraine treatment. If they do choose to participate, the patients will be brought to the angiography suite and transferred to the angiogram table. The patient will be prepped and draped in standard fashion for an angiogram and given instructions regarding the procedure for the day. The patient will receive local lidocaine at their groin site to minimize discomfort during standard arterial access for the purposes of the angiogram. Catheterization will commence into the external carotid artery. At this time, the patient's headache history will guide the decision for first vessel cannulation. If the patient has frontal migraines, the internal maxillary artery will be cannulated, for parietal headaches the focus will be on the superficial temporal artery, and the occipital artery for posterior, occipitally located symptoms, all on the side of the patient's migraines. A microcatheter will be placed at the origin of each respective artery and a control contrast injection will be performed to determine baseline vessel caliber and blood flow. Patients will be asked at this time if they are experiencing any pain or discomfort. If none, nitroglycerin will be drawn up and injected at a volume of 200µg diluted in 10ml saline into these vessels only. This is a standard injection dose for vasodilation for this medication and it is routinely available and used to treat vasospasm, or vasoconstriction that occurs after subarachnoid hemorrhage in the angiography suite. This dose has also been used in several cranial and cardiac studies and has not been association with adverse reactions related to systemic spread. The expectation is that this small dose will not reach systemic circulation. After 5 minutes, another contrast run will be performed to determine any change in vessel size and the patient will be questioned about any headache symptoms. After another 5 minutes, another contrast run will be performed to see if the nitroglycerin is still effective. If the patient describes no symptoms, the focus will be shifted to one of the other 2 external carotid artery branches to test them for the induction of headaches using the same nitroglycerin protocol. Each vessel will be evaluated for a full 10 minutes and if no vessel causes headache pain, the study will be terminated after a final control injection and femoral sheath removal. Pressure on the groin will be held for 20 minutes and the patient will be taken to the recovery room and monitored lying flat, as in standard fashion for 5 hours before being discharged home in order to prevent groin hematoma. They will again be evaluated for headaches or pain hourly until discharge, and be given another headache log to complete prior to their 2 week follow-up visit. The headache log will be collected at that time and this will complete the study for the patient.

If any vessel immediately, or with time produces headache pain, the patient will be queried regarding the type and quality of the headache, and asked if it is similar to their migraines. A 10 minute angiogram will be repeated at the vessel evaluated. With persistent headaches, a microballoon will be brought to the vessel origin, and it will be inflated to block flow in this vessel for 5 minutes before being deflated. As stated previously, there is no risk to occlusion of these vessels permanently, and certainly not temporarily as will be performed as part of this protocol. These non-critical vessels have dense anastomotic networks and are safe to occlude. Symptoms will be evaluated to see if any subside as a result of their occlusion. Five minutes after the balloon is deflated, another contrast run will be performed to evaluate the caliber of the studied vessel. After this run, the groin sheath will be removed and the above protocol will be followed until outpatient follow-up. If headache symptoms do not subside, the patient will be administered standard pain medication, fentanyl, which is given routinely during angiography at a dose of 25mcg to abate their pain. This is a low, tolerable, and safe dose that will be given with the assistance of our anesthesia colleagues, if necessary. Their headache pain will be closely monitored during the 5 hour recovery period, and given 1 more 25mcg dose during this period in order to fully subside any pain the patient still may have.

This angiogram will take approximately 30 minutes to complete, and it is a low risk procedure.. The vessels studied diagnostically will be solely extracranial and completely separate from intracranial vessels. Any anomalous communication identified between extracranial and intracranial vessels will automatically disqualify a patient from participation in this study.

Despite some minor discomfort from the groin puncture for the patient, with the assistance of an anesthesiologist the pain intra- and post-procedurally experienced by patients will be well controlled. The patient may also opt to receive the rescue pain medication at any time during the angiogram and discontinue the study.

As stated previously, the extracranial vascular circulation has a large anastomotic network such that a single vessel sacrifice can be performed without great risk. These vessels are sacrificed without sequelae intraoperatively routinely when performing craniotomies. In cases where a provocative artery can be found, occlusion of that vessel can lead to improved symptoms, as tested by temporary balloon occlusion without great risk. It is the hope that this pilot work to guide future interventions to control blood flow in these offending vessels, to see if migraines abate permanently with vessel removal from circulation. If these hypotheses are correct, interventions may be created to minimize patient's need for medication, improve their quality of life, and free them from the debilitation of their migraines.

ELIGIBILITY:
Inclusion Criteria:

* No changes to neurological exam within the preceding 6 months
* Requirement of a diagnostic cerebral angiogram for a previously treated aneurysm or arteriovenous malformation with no history of persistent disease
* A documented diagnosis of migraine made by a neurologist
* Migraines that are refractory to standard migraine pharmacologic treatment, with or without aura, either prophylactic or abortive, with persistent severe, debilitating symptoms
* Experience migraine symptoms at least twice a month
* Migraines symptomology which is discernible from other non-migraine headache pain
* Subjects must sign a consent form for both angiography and for participation in this study, and must be willing to undergo angiography for the evaluation of their symptoms

Exclusion Criteria:

* Patients with persistent intracranial vascular anomalies, such as aneurysms, which remain untreated, in whole or in part
* Patients taking vasoactive drugs including epinephrine, norepinephrine, dopamine, dobutamine, isoprenaline, dopexamine, milrinone, amrinon, levosimendan, glucagon, phenylephrine, metaraminol, ephedrine, vasopressin, digoxin, and levothyroxine
* Patients with underlying cardiac pathology including but not limited to coronary artery disease, heart attacks, or severe atherosclerosis
* Patients taking medications such as phosphodiesterase 5 (PDE5) inhibitors or other nitroglycerin analogues
* Patients with pulmonary disease requiring supplemental oxygen therapy
* Patients with contraindications to nitroglycerin or calcium channel blocker use
* Patients who have had coffee, tea, or alcohol in the 12 hours before the start of the angiogram
* Patients having other headache conditions, pain syndromes, or prior intracranial therapies or craniotomies for management of any vascular lesions that would require angiography for surveillance and confound their evaluation of their migraine pain
* Patients in whom the angiography demonstrates the anatomy is not appropriate for endovascular treatment, due to conditions such as:

  * Severe vessel tortuosity or stenosis
  * Vasospasm not responsive to medical therapy
  * Abnormal communication between intracranial and extracranial vessels either in the past or during the study procedure
* Patients who are not able to reliably report symptoms
* Patients without the capacity to consent
* Patients who do not consent to participate
* Patients who are pregnant
* Children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Migraine | 10 minutes
  The reporting of migraine-like pain after nitroglycerin administration

SECONDARY OUTCOMES:
Migraine log pre-procedure: severity measure | 2 weeks
  Severity of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: frequency measure | 2 weeks
  Frequency of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: quality measure | 2 weeks
  Quality of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: location measure | 2 weeks
  Location of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: alleviating factor measure | 2 weeks
  Alleviating factors of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: aggravating factor measure | 2 weeks
  Aggravating factors of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: associated symptom measure | 2 weeks
  Associated symptoms of migraines for 2 weeks prior to angiogram
Migraine log pre-procedure: therapies utilized measure | 2 weeks
  Therapies utilized for migraines for 2 weeks prior to angiogram
Artery dilation | 10 minutes
  Enlargement of the diameter of the vessel of interest after nitroglycerin administration
Migraine pain relief | 20 minutes
  Relief of induced migraine pain with temporary balloon occlusion of the dilated artery. Standard pain medication will also be available for treatment
Adverse reactions | 6 hours
  Monitoring for retroperitoneal hematoma, vascular injury, infection, contrast reaction, worsening contralateral headache symptoms, new neurologic deficit peri-procedurally until discharge
Migraine log follow-up post-procedure: severity measure | 2 weeks
  Severity of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: frequency measure | 2 weeks
  Frequency of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: quality measure | 2 weeks
  Quality of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: location measure | 2 weeks
  Location of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: alleviating factors measure | 2 weeks
  Alleviating factors of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: aggravating factor measure | 2 weeks
  Aggravating factors of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: associated factor measure | 2 weeks
  Associated symptoms of migraines for 2 weeks post-angiogram
Migraine log follow-up post-procedure: therapies utilized measure | 2 weeks
  Therapies utilized for 2 weeks after angiogram until follow-up clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: David J Altschul, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoenen J. Hypoxia, a turning point in migraine pathogenesis? Brain. 2016 Mar;139(Pt 3):644-7. doi: 10.1093/brain/awv402. No abstract available. PMID 26917583
- [Background] Stoeckelhuber BM, Suttmann I, Stoeckelhuber M, Kueffer G. Comparison of the vasodilating effect of nitroglycerin, verapamil, and tolazoline in hand angiography. J Vasc Interv Radiol. 2003 Jun;14(6):749-54. doi: 10.1097/01.rvi.0000079984.80153.5e. PMID 12817042
- [Background] Maruhashi T, Soga J, Fujimura N, Idei N, Mikami S, Iwamoto Y, Kajikawa M, Matsumoto T, Hidaka T, Kihara Y, Chayama K, Noma K, Nakashima A, Goto C, Higashi Y. Nitroglycerine-induced vasodilation for assessment of vascular function: a comparison with flow-mediated vasodilation. Arterioscler Thromb Vasc Biol. 2013 Jun;33(6):1401-8. doi: 10.1161/ATVBAHA.112.300934. Epub 2013 Mar 21. PMID 23520168
- [Background] McNiff EF, Yacobi A, Young-Chang FM, Golden LH, Goldfarb A, Fung HL. Nitroglycerin pharmacokinetics after intravenous infusion in normal subjects. J Pharm Sci. 1981 Sep;70(9):1054-8. doi: 10.1002/jps.2600700923. PMID 6101155
- [Background] Ferrari MD. The economic burden of migraine to society. Pharmacoeconomics. 1998 Jun;13(6):667-76. doi: 10.2165/00019053-199813060-00003. PMID 10179702
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Goadsby PJ, Charbit AR, Andreou AP, Akerman S, Holland PR. Neurobiology of migraine. Neuroscience. 2009 Jun 30;161(2):327-41. doi: 10.1016/j.neuroscience.2009.03.019. Epub 2009 Mar 19. PMID 19303917
- [Background] Costa C, Tozzi A, Rainero I, Cupini LM, Calabresi P, Ayata C, Sarchielli P. Cortical spreading depression as a target for anti-migraine agents. J Headache Pain. 2013 Jul 23;14(1):62. doi: 10.1186/1129-2377-14-62. PMID 23879550
- [Background] Evans RW. Diagnostic testing for migraine and other primary headaches. Neurol Clin. 2009 May;27(2):393-415. doi: 10.1016/j.ncl.2008.11.009. PMID 19289222
- [Background] Schoonman GG, van der Grond J, Kortmann C, van der Geest RJ, Terwindt GM, Ferrari MD. Migraine headache is not associated with cerebral or meningeal vasodilatation--a 3T magnetic resonance angiography study. Brain. 2008 Aug;131(Pt 8):2192-200. doi: 10.1093/brain/awn094. Epub 2008 May 23. PMID 18502781
- [Background] Nagata E, Moriguchi H, Takizawa S, Horie T, Yanagimachi N, Takagi S. The middle meningial artery during a migraine attack: 3T magnetic resonance angiography study. Intern Med. 2009;48(24):2133-5. doi: 10.2169/internalmedicine.48.2565. PMID 20009407
- [Background] Asghar MS, Hansen AE, Kapijimpanga T, van der Geest RJ, van der Koning P, Larsson HB, Olesen J, Ashina M. Dilation by CGRP of middle meningeal artery and reversal by sumatriptan in normal volunteers. Neurology. 2010 Oct 26;75(17):1520-6. doi: 10.1212/WNL.0b013e3181f9626a. PMID 20975053
- [Background] Amin FM, Asghar MS, Hougaard A, Hansen AE, Larsen VA, de Koning PJ, Larsson HB, Olesen J, Ashina M. Magnetic resonance angiography of intracranial and extracranial arteries in patients with spontaneous migraine without aura: a cross-sectional study. Lancet Neurol. 2013 May;12(5):454-61. doi: 10.1016/S1474-4422(13)70067-X. Epub 2013 Apr 9. PMID 23578775
- [Background] Arngrim N, Schytz HW, Britze J, Amin FM, Vestergaard MB, Hougaard A, Wolfram F, de Koning PJ, Olsen KS, Secher NH, Larsson HB, Olesen J, Ashina M. Migraine induced by hypoxia: an MRI spectroscopy and angiography study. Brain. 2016 Mar;139(Pt 3):723-37. doi: 10.1093/brain/awv359. Epub 2015 Dec 16. PMID 26674653
- [Background] Olesen J. The role of nitric oxide (NO) in migraine, tension-type headache and cluster headache. Pharmacol Ther. 2008 Nov;120(2):157-71. doi: 10.1016/j.pharmthera.2008.08.003. Epub 2008 Aug 23. PMID 18789357
- [Background] Meents JE, Neeb L, Reuter U. TRPV1 in migraine pathophysiology. Trends Mol Med. 2010 Apr;16(4):153-9. doi: 10.1016/j.molmed.2010.02.004. Epub 2010 Mar 27. PMID 20347391
- [Background] Evans MS, Cheng X, Jeffry JA, Disney KE, Premkumar LS. Sumatriptan inhibits TRPV1 channels in trigeminal neurons. Headache. 2012 May;52(5):773-84. doi: 10.1111/j.1526-4610.2011.02053.x. Epub 2012 Jan 30. PMID 22289052
- [Background] Totaro R, De Matteis G, Marini C, Baldassarre M, Carolei A. Sumatriptan and cerebral blood flow velocity changes during migraine attacks. Headache. 1997 Nov-Dec;37(10):635-9. doi: 10.1046/j.1526-4610.1997.3710635.x. PMID 9439084
- [Background] Shevel E. The trigeminovascular system--quo vadis? Headache. 2009 May;49(5):785-6. doi: 10.1111/j.1526-4610.2009.01415.x. No abstract available. PMID 19456890
- [Background] Shevel E. The extracranial vascular theory of migraine: an artificial controversy. J Neural Transm (Vienna). 2011 Apr;118(4):525-30. doi: 10.1007/s00702-010-0517-1. Epub 2011 Jan 5. PMID 21207080
- [Background] Shevel E. The extracranial vascular theory of migraine--a great story confirmed by the facts. Headache. 2011 Mar;51(3):409-417. doi: 10.1111/j.1526-4610.2011.01844.x. PMID 21352215
- [Background] Beekman R, Nijssen PC, van Rooij WJ, Wijnalda D. Migraine with aura after intracranial endovascular procedures. Headache. 2001 Apr;41(4):410-3. doi: 10.1046/j.1526-4610.2001.111006410.x. PMID 11318889
- [Background] Choi KS, Lee JH, Yi HJ, Chun HJ, Lee YJ, Kim DW. Incidence and risk factors of postoperative headache after endovascular coil embolization of unruptured intracranial aneurysms. Acta Neurochir (Wien). 2014 Jul;156(7):1281-7. doi: 10.1007/s00701-014-2095-8. Epub 2014 May 7. PMID 24801821
- [Background] Amin FM, Hougaard A, Schytz HW, Asghar MS, Lundholm E, Parvaiz AI, de Koning PJ, Andersen MR, Larsson HB, Fahrenkrug J, Olesen J, Ashina M. Investigation of the pathophysiological mechanisms of migraine attacks induced by pituitary adenylate cyclase-activating polypeptide-38. Brain. 2014 Mar;137(Pt 3):779-94. doi: 10.1093/brain/awt369. Epub 2014 Feb 5. PMID 24501094
- [Background] Edvinsson L, Linde M. New drugs in migraine treatment and prophylaxis: telcagepant and topiramate. Lancet. 2010 Aug 21;376(9741):645-55. doi: 10.1016/S0140-6736(10)60323-6. Epub 2010 Apr 21. PMID 20416945
- [Background] Meents JE, Hoffmann J, Chaplan SR, Neeb L, Schuh-Hofer S, Wickenden A, Reuter U. Two TRPV1 receptor antagonists are effective in two different experimental models of migraine. J Headache Pain. 2015;16:57. doi: 10.1186/s10194-015-0539-z. Epub 2015 Jun 24. PMID 26109436
- [Background] Hazard E, Munakata J, Bigal ME, Rupnow MF, Lipton RB. The burden of migraine in the United States: current and emerging perspectives on disease management and economic analysis. Value Health. 2009 Jan-Feb;12(1):55-64. doi: 10.1111/j.1524-4733.2008.00404.x. Epub 2008 Jul 30. PMID 18671771
- [Background] Bashir A, Lipton RB, Ashina S, Ashina M. Migraine and structural changes in the brain: a systematic review and meta-analysis. Neurology. 2013 Oct 1;81(14):1260-8. doi: 10.1212/WNL.0b013e3182a6cb32. Epub 2013 Aug 28. PMID 23986301
- [Background] Starling AJ, Dodick DW. Best practices for patients with chronic migraine: burden, diagnosis, and management in primary care. Mayo Clin Proc. 2015 Mar;90(3):408-14. doi: 10.1016/j.mayocp.2015.01.010. PMID 25744118
- [Background] Turner-Bowker DM, Bayliss MS, Ware JE Jr, Kosinski M. Usefulness of the SF-8 Health Survey for comparing the impact of migraine and other conditions. Qual Life Res. 2003 Dec;12(8):1003-12. doi: 10.1023/a:1026179517081. PMID 14651418
- [Background] WOLFF HG, TUNIS MM, GOODELL H. Studies on headache; evidence of damage and changes in pain sensitivity in subjects with vascular headaches of the migraine type. AMA Arch Intern Med. 1953 Oct;92(4):478-84. doi: 10.1001/archinte.1953.00240220026006. No abstract available. PMID 13091465
- [Background] Yonekawa Y. [Operative neurosurgery: personal view and historical backgrounds (3). Anterior circulation--pterional approach]. No Shinkei Geka. 2007 Jul;35(7):703-18. Japanese. PMID 17633515
- [Background] Kent RB 3rd, Thomas L. Temporal artery biopsy. Am Surg. 1990 Jan;56(1):16-21. PMID 2403766
- [Background] Sasanuma J, Goto T, Ogayama H, Sasaki J, Watanabe K. [Clinical effect of nitroglycerin (GTN) on prevention of cerebral vasospasm]. No Shinkei Geka. 1991 Mar;19(3):227-32. Japanese. PMID 1903850
- [Background] Tanaka Y, Masuzawa T, Saito M, Yamada T, Ebihara A, Iwasa H, Mori S. Combined administration of Fasudil hydrochloride and nitroglycerin for treatment of cerebral vasospasm. Acta Neurochir Suppl. 2001;77:205-7. doi: 10.1007/978-3-7091-6232-3_43. No abstract available. PMID 11563287
- [Background] Zenteno M, Santos Franco J, Moscote-Salazar LR, Lee A. [Endovascular management of cavernous sinus dural fistulas]. Bol Asoc Med P R. 2014;106(1):17-24. Spanish. PMID 24791359
- [Background] Rho MH, Kim BM, Suh SH, Kim DJ, Kim DI. Initial experience with the new double-lumen scepter balloon catheter for treatment of wide-necked aneurysms. Korean J Radiol. 2013 Sep-Oct;14(5):832-40. doi: 10.3348/kjr.2013.14.5.832. Epub 2013 Aug 30. PMID 24043982
- [Background] Baron EP. Headache, cerebral aneurysms, and the use of triptans and ergot derivatives. Headache. 2015 May;55(5):739-47. doi: 10.1111/head.12562. Epub 2015 Apr 22. PMID 25903747